CLINICAL TRIAL: NCT04080609
Title: A Single Dose, Open Label, Drug-drug Interaction Study to Investigate the Pharmacokinetics and Safety of Dorzagliation Administered Alone or in Combination With Rifampicin in Healthy Subjects
Brief Title: DDI Study Between Dorzagliatin and Rifampicin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HMM0108
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Dorzagliatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential arm (Experimental): Dorzagliatin was administered single dose; after wash-out, rifampicin was dosed continuously for 9 days, with Dorzagliatin dosed simultaneously on day 8.
  Interventions: Drug: Dorzagliatin

INTERVENTIONS:
Drug: Dorzagliatin — GKA currently under clinical development

SUMMARY:
The purpose of this drug-drug interaction study is to investigate the impact of rifampicin on the pharmacokinetics of Dorzagliatin.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 50 kg (male) or ≥ 45 kg (female)
* BMI within 19～26 kg/m2

Exclusion Criteria:

* History or disease status that may impact the ADME of the study
* Use of any drugs, OTCs, or hebal within 4 weeks of screening
* Drug abuse
* Blood donation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 96 hours
  Peak plasma concentration
AUClast | up to 96 hours
  Area under the plasma concentration curve

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital of Xuhui District, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No